Laureate Institute for Brain Research, Inc., Tulsa, OK, United States

| RESEARCH SUBJECT INFORMATION AND CONSENT FORM | |
|---|---|
| TITLE: | Neural response to inflammatory challenge in major depressive |
| | disorder |

# After reading and discussing the information in this consent form you should know:

- Why this research study is being done;
- · What will happen during the study;
- Any possible benefits to you;
- The possible risks to you;
- Other options you could choose instead of being in this study;
- How your personal health information will be treated during the study and after the study is over;
- Whether being in this study could involve any cost to you; and
- What to do if you have problems or questions about this study.

Please read this consent form carefully.

#### RESEARCH SUBJECT INFORMATION AND CONSENT FORM

**TITLE:** Neural response to inflammatory challenge in major

depressive disorder

**PROTOCOL NO.:** 2020-004

WIRB® Protocol #20201159

**SPONSOR:** National Institute of Mental Health

**INVESTIGATOR:** Jonathan Savitz, PhD

6655 S Yale Ave

Tulsa, Oklahoma 74136

**United States** 

STUDY-RELATED

PHONE NUMBER(S): Jonathan Savitz, PhD

918-502-5155

918-481-4000 (24 hours)

#### RESEARCH CONSENT SUMMARY

You are being asked for your consent to take part in a research study. This document provides a summary of this research and describes the information that most people need to decide whether to take part in this research. Later sections of this document will provide all relevant details.

#### What should I know about this research?

- Someone will explain this research to you.
- Taking part in this research is voluntary. Whether you take part is up to you. If you do not take part or if you take part now and later drop out, it will not be held against you.
- If there is information you do not understand, ask questions and make sure your questions are answered before you decide if you will participate.

#### How long will I be in this research?

- Depressed participants: There are 10 study visits and we expect you to be in the study for about 6 months.
- Non-depressed participants: There are 4 study visits and we expect you to be in the study for about 10-21 days.

# Why is this research being done?

The purpose of this research is to understand how the immune system is altered in depression and how these changes in immunity may affect brain activity and symptoms of depression.

# What happens to me if I agree to take part in this research?

If you decide to take part in this research study, the general procedures include questionnaires, cognitive tests, MRI scans, blood draws, urine tests, an IV, EKGs, an infusion with lipopolysaccharide (LPS) or saline, and sleep measurements with wrist actigraphy (smart watch).

# Could being in this research hurt me?

The most important risks or discomforts that you may expect from taking part in this research include experiencing flu-like symptoms from the LPS infusion, discomfort during the blood draws and IV placement, and claustrophobia/anxiety during the MRI scans.

# Will being in this research benefit me?

It is not expected that you will personally benefit from this research; however, your participation should help us better understand how depression and stress affect the immune system, which may benefit others in the future.

#### **DETAILED RESEARCH CONSENT**

This consent form describes a research study. Research studies involve only individuals who choose to participate. Please take your time to make your decision about participating in the study.

This consent form may contain words that you do not understand. Please ask the Principal Investigator or the study staff to explain any words or information that you do not clearly understand. You may take home an unsigned copy of this consent form to think about or discuss with family or friends before making your decision.

# Why Have You Been Asked To Participate In This Study?

You are being asked to take part in this study because:

You are in good health

or

• You are in good health and have been diagnosed in the past with depression.

# Why Is This Study Being Done?

This project seeks to understand how the immune system is altered in depression and how these changes in immunity may affect brain activity and symptoms of depression. To do this we will use an investigational bacterial toxin that can initiate chemical reactions that are similar to those seen in individuals with mild sickness symptoms, such

as a slight increase in body temperature, muscle aches, or tiredness. It is a way of investigating the body's response to inflammation and how these changes may alter cognitive, emotional, or neural function. It has been given hundreds of times to healthy volunteers without any serious side effects.

# What Drugs and Devices Are Involved In This Study?

Lipopolysaccharide (LPS) is a component of the cell wall of bacteria such as *Escherichia coli (E. coli)*. Our immune systems recognize this sugar molecule and begin an inflammatory response to fight what "it thinks" is an infection. You will not be receiving live bacteria but rather these sugar molecules that activate/stimulate the immune system into launching an inflammatory response. You have a 2 in 3 chance of receiving LPS and a 1 in 3 chance of receiving saline (purified salt water) which will not cause any immune response.

The Magnetic Resonance Imaging (MRI - use of a magnetic field to produce an image) scanner is used to look at brain function and anatomy. The Laureate Institute of Brain Research (LIBR) is using the MRI scanner in a research (experimental) mode. U.S. Food and Drug Administration (FDA) approval has not been obtained for the particular ways that information about inter-personal interaction from the MRI may be used in this research; however, the MRI scanner will not be used for purposes outside its intended application. It is considered to be a non-significant risk investigational device.

A physiological recording system will also be used to monitor heart rate and breathing.

#### **How Many Subjects Will Take Part In The Study?**

About 200 subjects will take part in this study at the Laureate Institute for Brain Research (LIBR).

# What Is Involved In The Study?

The study involves:

- Questionnaires
- Laboratory tests
- Electrocardiogram (EKG)
- Physical Exam
- LPS injection or placebo (saline)
- An IV (Intravenous line)
- Blood draws
- Cognitive tests
- MRI scanning
- Physical Measurements

- Wrist actigraphy (a sensor unit used to measure gross motor activity such as a watch)
- Urine tests
- Meals and/or snacks
- Post Study Visits

Visit Schedule Summary:

# Visit 1

Visit 1 will take approximately 4 hours to complete. You will be consented to the study, have your blood drawn, receive a physical exam and an electrocardiogram (EKG), complete an hour-long MRI scan, and complete some questionnaires.

The blood draw at this visit will include testing for Hepatitis C and HIV. State/Provincial law requires positive test results for certain communicable diseases, including HIV, hepatitis, sexually transmitted infections, and tuberculosis, to be reported to a local health agency. Some of the tests for this study must be reported when positive. The study doctor can discuss this with you.

# Visit 2

| Timeline | LPS<br>or<br>Saline | EKG | Vital Signs | SARS<br>CoV-<br>2 | Urine<br>Screen &<br>Breathalyzer | Mood<br>Ratings | MRI | Cognitive<br>Testing | Blood<br>Draw | Physical<br>Symptoms<br>Scale | Lunch<br>or<br>Snack | MD<br>Discharge<br>Assessment |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 8:30 AM | | | | | | | | | | | | |
| 9:00 AM | | | | | | | | | | | | |
| 9:30 AM | | | | | | | | | | | | |
| 10:00 AM | | | | | | | | | | | | |
| 10:30 AM | | | | | | | | | | | | |
| 11:00 AM | | | | | | | | | | | | |
| 11:30 AM | | | | | | | | | | | | |
| 12:00 AM | | | | | | | | | | | | |
| 12:30 AM | | | | | | | | | | | | |
| 1:00 PM | | | | | | | | | | | | |
| 1:30 PM | | | | | | | | | | | | |
| 2:00 PM | | | | | | | | | | | | |
| 2:30 PM | | | | | | | | | | | | |
| 3:00 PM | | | | | | | | | | | | |
| 3:30 PM | | | | | | | | | | | | |
| 4:00 PM | | | | | | | | | | | | |
| 4:30 PM | | | | | | | | | | | | |
| 5:00 PM | | | | | | | | | | | | |

#### ALL TIMES ARE APPROXIMATE

#### Post Study Visits

There is a post infusion visit 1 day (visit 3) and at 1 week (visit 4) after your study visit 2. Each visit will last approximately 60 minutes. You will be asked questions about physical symptoms, depressive symptoms, and sleep quality. You will complete various questionnaires to obtain this information. There is a blood draw at each of these visits.

After the 1-week visit (visit 4), we will do a six-month follow-up for depressed participants, only. These visits will require completion of questionnaires by internet (mobile assessment) on four occasions, 2 in-person assessments (at 3 months and 6 months) which involve blood draws, questionnaires and clinical interviews, and three sets of sleep assessment, each lasting two weeks. For the sleep assessments, you will complete a short diary (5 mins) every night for two weeks and wear a wrist actigraph (smart watch) during these two-week periods.

#### Questionnaires

These tests and questionnaires about your health, mood, and personality will measure your mental and physical states.

# Laboratory Tests

You will have blood tests. A trained nurse will take a small amount of blood from a vein in your arm. Blood will be collected using sterile techniques by a person experienced in drawing blood. Blood will be drawn through a needle in your arm during Visit 1. Visit 2 has five blood draws so a peripheral intravenous (IVP) line will be placed in both arms. This is a small flexible catheter in the vein that blood can be taken from and the injection can be given. You will not be charged for any of these tests. We may give you up to 500 ml of normal saline in your IVP to help hydrate you. The blood will be used for the measurement of various immune markers, metabolic panels, and for genetic analysis.

| | | | # TBSP of blood |
|---------------|---------------|----------------|-----------------|
| Visit | # Blood Tubes | # ml of Blood* | * |
| Study visit 1 | 7 | 46 | 3 |
| Study visit 2 | 25 | 220 | 15 |
| Study visit 3 | 5 | 44 | 3 |
| Study visit 4 | 5 | 44 | 3 |
| Study visit 7 | 5 | 44 | 3 |
| Study visit | | | |
| 10 | 5 | 44 | 3 |
| Total for All | 52 | 442 | 30 |

\*approximately \*approximately

# Lipopolysaccharide (LPS) Injection

You will be given an intravenous injection of a low dose LPS or a placebo of normal saline by a Registered Nurse. Whether you receive LPS or a placebo is decided randomly (by chance). Two out of three participants will receive LPS and one out of three will receive saline. However, neither you nor your study doctor will know when you will receive the LPS or saline.

# MRI Scanning

You will be asked to participate in the MRI scanning. For your safety, you will be given a brief pre-screening form to complete. It will tell us if you have any metal inside your body. The pre-screening form may identify some unanticipated medical findings that prevent you from participating in the MRI scan. If so, these findings will remain as confidential as possible, and will be discussed with you by a researcher involved in this study. Female participants will have an over-the-counter urine pregnancy test immediately before the scanning session. You will not be allowed to participate in the study if the pregnancy test reads positive.

Prior to your scan, you will be taught some tasks for use in the scanner. This will take about 5 minutes. The tasks will be decision making tasks and you will have the opportunity to be paid up to \$30 during these tasks. See section below entitled "Will I be Paid for Participating in this Study?" for further information.

The MRI scanner rapidly takes pictures of your brain without exposure to radiation. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. During the MRI, you will lie on a table that can slide in and out of the cylinder. You will be asked to lie still during scanning by remaining as relaxed as possible. While in the scanner you will hear loud knocking noises, and you will be fitted with earplugs to muffle the sound. You will be able to communicate with the MRI staff at all times during your scan, and you may ask to be moved out of the machine at any time. We may also monitor your heart rate and respiration using a device on your finger and a rubber belt that fits loosely around your chest using the built-in scanner equipment.

The study will use anatomical MRI and functional Magnetic Resonance Imaging (fMRI). During the fMRI, the MRI scanner measures changes in blood oxygen levels in different neuroanatomical regions while you perform mental tasks. This procedure involves *no* injections or radiation and will provide us with information about which neuroanatomical areas become more active (that is, receive more blood oxygen) while you are performing the tasks.

There will be two brain-scanning sessions (one at visit 1 and one at visit 2). The time in the scanner will be approximately 1 hour for each scan.

#### Physical Measurements

Your weight, height, blood pressure, pulse, Electrocardiogram (EKG), breathalyzer, and other like measurements will be obtained for research purposes.

#### **Urine Tests**

If you are a female of childbearing years, you will receive an over-the-counter urine pregnancy test during the screening visit and prior to the LPS/saline administration.

# Meals and/or Snacks

During Visit 2, you will be provided with meals and or snacks as needed.

# Wrist actigraphy

You may be asked to wear a small device on your wrist that is about the size of a wristwatch. This device will record your physical activity during the day and sleep quality at night. You will be asked to wear the watch both at night and during the day until the end of the sleep assessment or two weeks. In addition, you will be asked to complete a sleep diary about each night of sleep.

#### How Long Will You Be In The Study?

For depressed participants, there are 10 study visits. We expect you will be in this study for up to 28 weeks.

For non-depressed participants, there are 4 study visits. We expect you will be in this study for 10-21 days.

There may be circumstances under which your participation in the study may be stopped by the investigator without your consent. Functional MRI is dependent upon measuring very small changes in blood flow in the brain. Therefore, there may be times in which the information collected will be unusable due either to a scanner malfunction or from you moving your head too much. Under these circumstances your participation may be stopped without your consent.

You may stop participating in this study at any time. You may also refuse to be contacted again in the future about participating in the study again.

# What Are The Risks Of The Study?

#### Questionnaires

There is no medical risk associated with the questionnaires. You may experience temporary discomfort, including anxiety and sadness, when recalling particularly negative memories. Members of the research staff are trained to help you if you have an unusually strong reaction to these memories. You can also stop the procedure at any time. Also, if you show a strong reaction, such as extreme sadness, to any part of the study, researchers will stop the procedure and help you relax before leaving the LIBR.

#### **Blood Collection**

For the blood collections, you may have some discomfort and bruising at the site of needle entry. There is a small risk of fainting or infection in the area of the needle insertion.

# LPS injection

Although we will be administering low doses of LPS, you may experience some side effects, such as an increase in body temperature, decreased or increased heart rate, increased or decreased blood pressure, nausea, shivering, headache, muscle pain, fatigue and an increase in symptoms of anxiety and depression. In rare cases (~1%), there is a possibility of vomiting or diarrhea.

Some significant changes in heart rate/blood pressure and body temperature have been found to occur following LPS administration, although such abnormalities are only found at doses that are 4-fold greater than the highest dose used in this study. There also is one recorded case of asystole (a state of no electrical activity from the heart, potentially leading to cardiac arrest) in a participant who was thought to be dehydrated and who received more than double the dose of LPS that you will be receiving in this study.

Throughout the infusion protocol and for several hours following infusion, you will be carefully monitored with repeated vital signs and behavioral observations. If you do show any of the symptoms listed here, they will be most prominent for two to three hours after the LPS dose and then lessen by six hours after the dose is given. If any symptoms are particularly distressing, they can be relieved by aspirin, ibuprofen or acetaminophen. If you do show a clinically significant increase in physical symptoms or depressive symptoms, the study physician will be called and will evaluate you to determine the severity of your symptoms. If there are significant symptoms, the study physician will continue to monitor you until the symptoms are resolved and will not discharge you from LIBR until symptoms have returned to normal.

There is also a risk that you may become more depressed during the study. Therefore, we will follow-up with 2 in-person visits, one day and one week after visit 2. The study physician will be available for you to contact if you continue to experience a worsening of depressive symptoms after the study is completed.

Common risks and complications (more than 5%; > 1/20 individuals):

- Physical symptoms (chills, body aches, headache, and nausea)
- Increased temperature (increase of less than 2 degrees; ~100° F)
- Increased heart rate
- Increased fatique

Rare risks and complications (1%; 1 person in 100)

- Significant reduction in blood pressure
- Vomiting
- Diarrhea

An MD and RN will be available during the study visit to monitor you for any problems.

# Frequently Asked Questions about LPS

Question: Is the E. coli bacteria that will be used in the study alive?

**Answer:** No. When we expose you to E. coli, we are actually exposing you to a part of the cell wall of the E. coli bacteria. The cell wall of the bacteria stimulates your immune system to send out immune agents to clear it from your system. So, you will only be exposed to a specific part of the bacteria that has been isolated and that is known to induce an immune response by your body.

**Question:** How can this study be safe when I keep hearing that E. coli can make you very sick?

Answer: First, when you get E. coli from food (which is what can make people sick), you are getting the whole bacteria into your gut and bloodstream. When we expose you to E. coli here, we are exposing you to only a part of the E. coli bacteria – the cell wall. Moreover, the E. coli that we use in this study is the same kind of E. coli that is found naturally in your gut, whereas the kind of E. coli that you can be exposed to from food can be one of several different types of E. coli that your body may not be as familiar with. Second, we will be giving you a very low dose of LPS that is tightly controlled and is known to elicit very few sickness symptoms. This type of E. coli cell wall has been used in many different studies to better understand the immune system and over 3000 people have been exposed to it with no negative consequences. When you are exposed to E. coli in your food, you are being exposed to it in much larger doses that are obviously not controlled.

**Question:** How long will the E. coli cell wall be in my system?

**Answer:** The cell wall of the E. coli will actually be completely degraded and destroyed within 15 minutes of it entering your body. All of the possible symptoms that occur in response to e. coli exposure (aches, fatigue, nausea) are the result of the immune system sending out signals to your brain to engage in certain behaviors to recover from this foreign agent. We are interested in these symptoms that occur in response to exposure to E. coli cell wall.

**Question:** What if I have a bad reaction to the E. coli cell wall?

**Answer:** If you find that the symptoms that occur in response to E. coli cell wall exposure are too distressing or uncomfortable, we can resolve many of these symptoms by having you take aspirin, ibuprofen or acetaminophen. This should reduce fever and any aches, pains, or chills that accompany E. coli cell wall exposure. In addition, you will have the attention of the nurses and doctors at LIBR, who can provide full medical services to you to help resolve any unwanted or distressing symptoms.

**Question:** How long will it take for my body to go back to normal?

**Answer:** As mentioned previously, the E. coli cell wall will be completely out of your system within about 15 minutes. The symptoms that you may experience in response to the e. coli cell wall, however, will last longer. Symptoms such as fatigue, aches, nausea, and chills will peak at around 1-2 hours after E. coli cell wall exposure. After this time, they should continue to decrease. For most individuals, all symptoms will be gone within 6 hours after exposure to E. coli cell wall.

#### <u>Brain MRI</u>

People are at risk for injury from the MRI magnet if they have any of the following metal implants or fragments:

- pacemakers or other implanted electronic devices
- brain stimulators
- dental implants
- aneurysm clips (metal clips on the wall of a large artery)
- metallic prostheses (including metal pins and rods, heart valves, and cochlear implants)
- permanent eyeliner
- implanted delivery pump
- shrapnel fragments

Welders and metal workers are also at risk for injury because they may be unaware of small metal fragments in the eye.

You will be screened for these implants or metal fragments before the study, and if you have any of them, you will not receive an MRI scan and cannot be in the study. Tell the study doctor if you are uncertain whether you have any metal objects in your body. In addition, all magnetic objects (for example, watches, coins, jewelry, and credit cards) must be removed before entering the MRI scanner room.

Because of potential risk to an unborn baby, women who are pregnant are excluded from having an MRI and cannot be in the study.

You will be asked to complete an MRI screening form and to sign a separate MRI consent form for each MRI scan.

There are no known long-term risks or consequences of MRI scans. However, you may become uncomfortable because you will be lying in a small space. Some people are bothered by the loud thumping noises made by the scanner. You will wear earplugs to reduce the noise and increase your comfort during scanning. LIBR study staff will closely and continuously monitor you throughout the scanning procedure. You will be removed from the scanner immediately if you request to be removed.

# Physical Measurements

There are no known risks in taking your physical measurements.

#### Genetic Testing

A Federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information.

This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when making a decision to hire, promote, or fire you or when setting the terms of your employment.

Be aware that GINA does not protect you or your family against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Also, GINA does not prohibit discrimination of individuals with a genetic disorder that has been diagnosed. However, in order to do everything possible to keep this from happening, the results of this test along with information that could identify you (as described in the next paragraph) will only be shared with the study staff. This means that the genetic information we obtain will not be made available to you, your family

members, your private physician, your employer, your insurance company or any other party as allowed by law.

#### Delaying Treatment

You may participate in this study if you are currently unmedicated or if you are currently receiving anti-depressant treatment. You will not be asked to discontinue any medications you have previously been taking for the purposes of this study. It is very important that you inform the principal investigator or his assistant of your recent medication use. You should also check with the study doctor or his assistant before taking any over-the-counter or prescribed medications while you are in the study. We request this communication in order to be certain that you do not take any medication that might interfere with the study measurements, interpretation of the findings, or may cause side effects. It is also important that you do not make major changes to your routine before or during the study — e.g. start an exercise program.

If you are unmedicated, in order to avoid long delays in treatment for conditions that might require you to take medications, you will be provided an opportunity to participate in the study within two weeks of the signing of this consent form. You should not participate in this study if it will be difficult for you to delay treatment longer than two weeks. To reduce the risks associated with delaying treatment, during this drug-free period, you may contact the study doctor. The study doctor will put you in touch with a healthcare professional with whom you can consult.

If you are unmedicated, the risks of delaying treatment may include a worsening of your symptoms of depression and the development of suicidal thoughts. Suicide is a risk of uncontrolled depression. You should notify the study doctor immediately if you have suicidal thoughts.

There is the possibility of hospitalization or a stop in your participation by the principal investigator in the study if it becomes clear that continued participation is not in your best medical interest.

# Pregnancy Risks

If you are a woman of child-bearing years, you must not be pregnant while participating in this study. There may be other risks from study participation that currently are unknown.

# You Should NOT Participate in the Study if:

- You are pregnant or suspect that you may be pregnant
- You have heart disease, kidney disease or another chronic medical illness.
- You have a chronic infectious illness or an autoimmune disease
- You have had a recent infection (e.g. cold or flu) or were vaccinated in the last 2 weeks

- You are feeling suicidal
- You are currently using hormone-containing medications (except contraceptives)
- You are currently taking pain medications
- You are currently taking medications for your heart
- You are claustrophobic

There may be unknown risks associated with this study.

# Are There Benefits To Taking Part In The Study?

There is no direct medical benefit anticipated for you in this study. Your participation should help us better understand how depression and stress affect the immune system.

# What Are The Costs Of Participating In The Study?

Neither you nor your health insurance will be charged for any of the study tests, procedures, or activities. If you need to be hospitalized, voluntarily or involuntarily, LIBR does not intend to provide payment for this, and you or your insurance provider will be billed for these costs.

# Will You Be Paid For Participating In This Study?

| | Approximate Time in | _ | Incentive |
|---|---|---|---|
| Visit 1 | Hours | Compensation | Earned |
| Consent | 0.5 | | |
| Blood draw, Physiological measures & EKG | 0.5 | \$25 | |
| Interviews & behavioral evaluations | 2 | \$20 | |
| MRI scan | 1 | \$50 | |
| Incentive Tasks in scanner | 0 | | up to \$30 |
| Total for Visit 1 | 4 | \$95 | up to \$125 |
| Visit 2 | | | |
| Blood draw x5, Physiological measures & EKG x2 | 1 | \$25 | |
| IV placement x2 | 0.5 | \$50 | |
| Interviews & behavioral evaluations x5 | 4 | \$40 | |
| LPS or Placebo injection | 2 | \$100 | |
| Lunch & Rest provided | 1 | \$0 | |
| MRI scan | 1 | \$50 | |
| Incentive Tasks in scanner | | | up to \$30 |
| Total for Visit 2 | 9.5 | \$265 | up to \$295 |
| Visits 3 and 4 (x2) | | | |
| Blood draw | 0.5 | \$25 | |
| Interviews & behavioral evaluations | 0.5 | \$20 | |

| Total per Visit | | \$45 |
|------------------------------------------|-----|-------|
| Total for visits 3 and 4 | | \$90 |
| Visits 5, 6, 8 and 9 (mobile assessment) | | |
| Internet questionnaires | 0.5 | \$20 |
| Total for visits 5,6,8 and 9 | | \$80 |
| Visits 7 and 10 (3 month and 6 month in | | |
| person assessments) | 1.5 | \$60 |
| Blood draws | 0.5 | \$25 |
| Total for visits 7 and 10 | | \$170 |

| Mobile sleep assessment | | |
|----------------------------------|-----------|-------|
| Sleep diary and wrist actigraphy | (2 weeks) | \$100 |
| Total for sleep assessments | | \$300 |

You will be paid through a ClinCard (similar to a debit card) that may be used approximately 1 business day after the visit.

# What Other Options Are There?

This study is for research purposes only, so your other option is not to participate in the study. You may still be treated for your symptoms without being in the study.

# Confidentiality

#### What information may be used and given to others?

The study doctor will get your personal and medical information. For example:

- Past and present medical records
- Research records
- Records about phone calls made as part of this research
- · Records about your study visits.

# THE INFORMATION AUTHORIZED FOR RELEASE MAY INCLUDE RECORDS WHICH MAY INDICATE THE PRESENCE OF A COMMUNICABLE OR NONCOMMUNICABLE DISEASE.

This information is made confidential by law and can be released only with your permission except by order of the court or health department in certain limited cases of persons who have risk of exposure of the diseases. Information from this study may be submitted to governmental agencies in other countries where the study medication may be considered for approval. Because of the need to release information to these parties, absolute confidentiality cannot be guaranteed.

# Who may use and give out information about you?

The study doctor and the study staff.

# Who might get this information?

The sponsor of this research. "Sponsor" means any persons or companies that are:

- working for or with the sponsor, or
- owned by the sponsor.

#### Your information may be given to:

- The U.S. Food and Drug Administration (FDA)
- Department of Health and Human Services (DHHS) agencies
- WCG Institutional Review Board (WCGIRB)

#### Why will this information be used and/or given to others?

- to do the research,
- to study the results, and
- to make sure that the research was done correctly
- State/Provincial law requires positive test results for certain communicable diseases to be reported to a local health agency. Some of the tests for this study must be reported when positive. The study doctor can discuss this with you.

If the results of this study are made public, information that identifies you will not be used.

#### **Databases**

Data from this study will be submitted to the National Institute of Mental Health Data Archive (NDA) at the National Institutes of Health (NIH). NDA is a large database where deidentified study data from many NIH studies are stored and managed. Deidentified study data means that all personal information about you (such as name, address, birthdate) is removed and replaced with a code. The code cannot be used to identify you and the study team will never send your personal information to the NDA.

Researchers across the world can request your deidentified study data for different research projects. Every researcher (and the institution to which they belong) who requests your deidentified study data must promise to keep your data safe and not to try to learn your identity. Experts at the NIH who know how to keep your data safe will review each request carefully to reduce risks to your privacy. Sharing your study data does have some risks, although these risks are rare. Your study data could be accidentally shared with an unauthorized person who may attempt to learn your identity.

The researchers will make every attempt to protect your identity. While you may not benefit directly from allowing your study data to be shared with NDA, sharing your deidentified study data helps researchers learn new and important things about brain science more quickly than before.

It is possible that you will participate in more than one study that sends data to NDA. NDA can connect your data from different studies by matching the code number on your deidentified data from each study. This data matching helps researchers who use NDA data to count you only one time.

You may decide now or later that you do not want your study data to be added to NDA. You can still participate in this research study even if you decide that you do not want your data to be added to NDA. If you know now that you do not want your data in NDA, please tell the study staff. If you decide any time after today that you do not want your data to be added to NDA, contact the study staff and they will tell NDA to stop sharing your study data. Once your data is part of NDA, the study researchers cannot take back the study data that was shared before they were notified that you changed your mind. If you would like more information about NDA, it is available on-line at <a href="http://nda.nih.gov">http://nda.nih.gov</a>.

# **Certificate of Confidentiality**

We will do everything we can to keep others from learning about your participation in this study. To further help us protect your privacy, we have obtained a Certificate of Confidentiality from the United States Department of Health and Human Services (DHHS). With this Certificate, we cannot be forced (for example by court order or subpoena) to disclose information that may identify you in any federal, state, local, civil, criminal, legislative, administrative, or other proceedings. The researchers will use the Certificate to resist any demands for information that would identify you, except to prevent serious harm to you or others, and as explained below.

You should understand that a Certificate of Confidentiality does not prevent you, or a member of your family, from voluntarily releasing information about yourself, or your involvement in this study.

If an insurer or employer learns about your participation, and obtains your consent to receive research information, then we may not use the Certificate of Confidentiality to withhold this information. This means that you and your family must also actively protect your own privacy. Disclosure will be necessary, however, upon request of DHHS for the purpose of audit or evaluation, and is limited only to DHHS employees involved in the review.

You should understand that we will in all cases, take the necessary action, including reporting to authorities, to prevent serious harm to yourself, children, or others. An example of a reportable incident would be child abuse or neglect.

# What if I decide not to give permission to use and give out my health information?

Then you will not be able to participate in this research study.

# May I review or copy my information?

Yes, but only after the research is over.

# May I withdraw or revoke (cancel) my permission?

Yes, but this permission will not stop automatically.

You may withdraw or take away your permission to use and disclose your health information at any time. You do this by sending written notice to the study doctor. If you withdraw your permission, you will not be able to stay in this study.

When you withdraw your permission, no new health information identifying you will be gathered after that date. Information that has already been gathered may still be used and given to others.

# Is my health information protected after it has been given to others?

There is a risk that your information will be given to others without your permission and may no longer be protected.

If you have any questions or concerns about your privacy rights, you should contact the LIBR Chief Operating Officer, Colleen McCallum at 918-502-5180 or via email at cmccallum@laureateinstitute.org.

You have the right to access the medical information that has been collected about you as a part of this research study. However, you may not have access to this medical information until the entire research study is finished.

#### What If You Are Injured While Participating In This Study?

If you get hurt or sick while participating in this study, emergency medical treatment is available from the Saint Francis Hospital and/or the Laureate Psychiatric Clinic and Hospital. If you get sick after the study is completed, call 911 in an emergency. Be sure to tell the emergency staff and other healthcare providers of your participation in this study. Contact the Principal Investigator of this study, Jonathan Savitz, PhD, as soon as possible at 918-502-5155 or 918-481-4000 (24 hours) if you think you have a research-related injury or illness.

You or your health insurance provider will be billed to cover the cost of the medical or emergency services provided. Some insurance carriers may not provide coverage for injuries received while participating in a research study. You are encouraged to contact

your insurance carrier to determine whether coverage is available. Otherwise, you may have unexpected expenses as a result of your participation in this study. No funds have been set aside by LIBR to compensate you if you are hurt or get sick. However, you still have the right to bring a lawsuit if you think you were harmed and deserve compensation.

You do not give up any of your legal rights by signing this consent form.

# Who Will Provide Funding For The Study?

Funding for this research study will be provided by the Laureate Institute for Brain Research and through a grant from the National Institute of Mental Health.

#### What Are Your Rights As A Participant?

Taking part in this study is voluntary. You may choose not to participate. Refusal to participate will involve no penalty or loss of benefits to which you are otherwise entitled. If you agree to participate and then decide against it, you can withdraw for any reason and leave the study at any time without penalty or loss of benefits to which you are otherwise entitled.

# Can The Researchers Remove Me From This Study?

The investigator may withdraw you from this research activity (without your consent) if certain circumstances arise. For example, you may be withdrawn from this study if the investigator feels that your continued participation places you at unnecessary risk or harm or you become ineligible (because of illness) to continue or because of non-adherence to protocol instructions. You may have to drop out, even if you would like to continue. The investigators will make a decision and let you know if it is possible for you to continue. The decision will be made to protect your health and safety.

# What If There Are New Findings?

We will provide you with any significant new findings developed during the research study that may affect your health, welfare, or willingness to continue your participation in this study. You may be asked to sign a new consent form if this occurs.

#### Whom Should You Call If You Have Questions Or Problems?

Your contact person for this study is Jonathan Savitz, PhD. He can be reached during business hours at 918-502-5155.

If you have questions about your participation in this study, concerns, or complaints about the study, or have a research-related injury, contact the study doctor, Jonathan Savitz, PhD, at 918-502-5155 or 918-481-4000 (24 hours). For emergencies call 911.

If you have questions about your rights as a research subject or if you have questions, concerns, input, or complaints about the research, you may contact:

WCG Institutional Review Board (WCG IRB)

Telephone: 855-818-2289

E-mail: researchquestions@wcgirb.com

WCGIRB is a group of people who perform independent review of research.

WCGIRB will not be able to answer some study-specific questions, such as questions about appointment times. However, you may contact WIRB if the research staff cannot be reached or if you wish to talk to someone other than the research staff.

Do not sign this consent form unless you have had a chance to ask questions and have received satisfactory answers to all of your questions.

If you agree to be in this study, you will be given a signed and dated copy of this consent form.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

IRB APPROVED AS MODIFIED Apr 29, 2024

Date

# **Signature**

I have read the information in this consent form. I have been given an opportunity to ask questions. All my questions about the study and my participation in it have been answered.

# I Agree To Participate In This Study

| I authorize the use and disclosure of my health information to the parties authorization section of this consent for the purposes described above. | s listed in the |
|---|---|
| PRINTED NAME OF PARTICIPANT | |
| Consent Signature | |
| PARTICIPANT SIGNATURE (18 years and older) | Date |
| I agree to deidentified data being shared with the NDA | |
| ☐ Yes | |
| □ No | |
| SIGNATURE OF PERSON CONDUCTING INFORMED CONSENT DISCUSSION | Date |
| ☐ The subject passed the LPS Consent Test with a score of 85% or mo | ore. |
| ☐ The subject did not pass the LPS Consent Test. | |

PRINTED NAME OF PERSON CONDUCTING THE

INFORMED CONSENT DISCUSSION